CLINICAL TRIAL: NCT01797523
Title: A Phase II, Single-Arm Study of RAD001 (Everolimus), Letrozole, and Metformin in Patients With Advanced or Recurrent Endometrial Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0543; NCI-2013-00960 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer; Advanced or Recurrent Endometrial Carcinoma; Metformin; Letrozole; Femara; Everolimus; Afinitor; Zortress; RAD001
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Metformin; Letrozole; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Letrozole + Metformin + RAD001 (Experimental): Patients have a 7-10 day lead in period where they take Metformin alone. The starting dose of Metformin 500 mg by mouth daily for 4 days and then increased to 500 mg by mouth twice a day. Everolimus and Letrozole added and considered the start of Cycle #1.
  Everolimus administered by mouth as once daily dose of 10 mg. Letrozole 2.5 mg tablet by mouth once daily. The oral dose of Everolimus should be taken together with the daily dose of Letrozole 2.5mg.
  Interventions: Drug: Metformin; Drug: Letrozole; Drug: Everolimus

INTERVENTIONS:
Drug: Metformin — 500 mg by mouth daily for 4 days on Days 1 - 4 of Cycle 0 and then 2 times a day (about 12 hours apart) every day after that. Metformin taken for 7 - 10 days in Cycle 0 before Cycle 1 begins.
Drug: Letrozole — 2.5 mg tablet by mouth once daily in a 28 day cycle.
  Other Names: Femara
Drug: Everolimus — 10 mg by mouth once daily in a 28 day cycle.
  Other Names: Afinitor; Zortress; RAD001

SUMMARY:
The goal of this clinical research study is to learn if the combination of everolimus, letrozole, and metformin can help to control recurrent or progressive endometrial cancer. The safety of this drug combination will also be studied.

Everolimus is designed to block a protein inside cancer cells that is involved in cancer growth.

Letrozole is designed to block a protein from making estrogen. This may interfere with the growth of cancer cells.

Metformin is commonly used to control blood sugar levels in patients with diabetes. It is designed to lower insulin levels, which may slow or stop the growth of endometrial cancer cells.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study and you are not already taking metformin, you will take metformin before you begin the regular study cycles (Cycles 1 and beyond). This will be called "Cycle 0." You will take metformin by mouth 1 time a day on Days 1-4 of Cycle 0 and then 2 times a day (about 12 hours apart) every day after that. You will take metformin for 7-10 days in Cycle 0 before Cycle 1 begins. If you are already taking metformin, you will continue your regular dose and start Day 1 of Cycle 1. If you are already taking metformin but your dose is less than 1000mg/day, your dose will be slowly raised up to the study dose over the course of 7-10 days and then you will start Cycle 1. In Cycles 1 and beyond, all participants will take all 3 drugs at a time. You should take metformin with food.

Starting in Cycle 1, you will take everolimus 1 time a day by mouth at about the same time every day. You should take it either consistently with food every day or consistently without food every day.

Starting in Cycle 1, you will take letrozole 1 time a day by mouth at about the same time every day.

It is very important for you to take the study drugs just as the study doctor tells you. Do not skip any doses unless your study doctor tells you to skip doses. If you throw up after taking the study drugs, you should NOT take another tablet that day. Let your study doctor know that you got sick. If you forget to take the study drugs one day, do not take any extra doses the next day. Call your study doctor and ask for advice.

There are 4 weeks in each cycle (except Cycle 0).

Study Visits:

Every cycle (+/- 10 days):

* You will have a physical exam, including measurement of your vital signs and weight.
* Your performance status will be recorded.
* You will be asked about any side effects you may have had.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* If the doctor thinks it is needed, blood (about 1 teaspoon) will be drawn to check for hepatitis.

After Cycles 2, 4, and 6 and then every 3 cycles after that (Cycles 9, 12, 15, and so on) (+/- 10 days):

* You will have scans such as a CT scan and/or MRI to check the status of the disease.
* If you have chest disease, you will have a CT scan of the chest.
* If the disease could be felt in the pelvis at the beginning of the study, you will have a pelvic exam

After every other cycle (Cycles 2, 4, and so on), blood (about 1 teaspoon) will be drawn for routine tests.

Length of Treatment:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

End-of-Treatment Visit:

Within 4 weeks after the last dose of study drugs:

* You will have a physical exam, including a pelvic exam and measurement of your vital signs and weight.
* Your performance status will be recorded.
* You will be asked about any side effects you may have had.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will have scans such as a CT scan and/or MRI to check the status of the disease.
* If you have chest disease, you will have a CT scan of the chest.

Follow-Up:

You will have follow-up visits as often as the doctor thinks is needed. At every visit:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* You will be asked about any side effects you may have had.
* If the doctor thinks it is needed, you will have scans such as a CT scan and/or MRI to check the status of the disease.
* If you have chest disease, you will have a CT scan of the chest.

As often as the doctor thinks is needed, the study staff will call you to ask about side effects you may have had. These calls should last 5-10 minutes.

.

This is an investigational study. Everolimus is FDA approved and commercially available to treat kidney, breast, and pancreatic cancers. Letrozole is FDA approved and commercially available to treat breast cancer and ovarian cancer. Metformin is FDA approved and commercially available to treat diabetes. The combination of everolimus, metformin, and letrozole in this study to treat endometrial cancer is investigational.

Up to 64 patients will be enrolled in this study. Up to 59 may take part at MD Anderson. Up to 5 patients per site may be enrolled at MD Anderson Cooper and Spartanburg Regional Healthcare System and Harris Health System.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically-confirmed advanced or recurrent endometrial carcinoma (endometrioid and mixed tumors, any grade) that is refractory to curative therapy or established treatments
2. Patients must have had no more than two prior chemotherapeutic regimens for recurrent management of endometrial carcinoma. Chemotherapy administered in conjunction with primary radiation as a radio-sensitizer is not counted as a prior treatment for recurrent or advanced disease
3. Prior radiation therapy of any kind is allowed
4. All patients must have measurable disease per RECIST 1.1 defined as at least one target lesion that can be accurately measured in at least one dimension (>/=10mm longest dimension to be recorded; Lymph nodes must be >/=15 mm per short axis). Each lesion must be > 20 mm when measured by palpation or conventional imaging techniques (CT or MRI - based on primary physician preference) or >10 mm with spiral CT scan. Measurable lesions must be at least 2 times the slice thickness in millimeters. Tumors within a previously irradiated field will be designated as non-target lesions unless progression is documented. Ascites and pleural effusions are not considered measurable disease. If the measurable disease is confined to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology
5. Patients must not be of child-bearing potential. Patients are considered not of child-bearing potential if they are surgically sterile (they have undergone a total hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal for greater than 12 months. Patients in whom ovaries are present and were not previously menopausal at the time of hysterectomy, should have a serum estradiol <10 pm/mL to confirm ovarian senescence.
6. Patients must be off all other anti-tumor therapies (including immunologic or hormonal agents) for at least four weeks prior to study registration.
7. Age >/= 18 years
8. GOG performance status </= 2
9. Adequate bone marrow function as shown by: ANC >/= 1.5 x 10^9/L, Platelets >/= 100 x 10^9/L, Hb >9 g/dL
10. Adequate liver function as shown by: a. serum bilirubin </= 1.5 x ULN b. ALT and AST </= 2.5x ULN (</= 5x ULN in patients with liver metastases); Adequate renal function:serum creatinine < 1.4mg/dL (per manufacturer, metformin is contraindicated in the presence of renal dysfunction defined as a serum creatinine> 1.4 mg/dL in females and in patients with abnormal clearance) ; Fasting serum cholesterol </= 240 mg/dL OR </=7.75 mmol/L AND fasting triglycerides </= 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication
11. Signed informed consent
12. Prior treatment with letrozole is allowed.

Exclusion Criteria:

1. Patients who have uterine sarcomas, carcinosarcomas, any serous histology or pure clear cell carcinomas
2. Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.)
3. Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
4. Prior treatment with any investigational drug within the preceding 4 weeks
5. Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed
6. Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period. Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
7. Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
8. Other malignancies within the past 3 years except for basal or squamous cell carcinomas of the skin.
9. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as: a. Symptomatic congestive heart failure of New York heart Association Class III or IV; b. Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease; c. Severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air; d. Active (acute or chronic) or uncontrolled severe infections
10. CONTINUED FROM 10 - e. Liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C). Note: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. HBV DNA and HCV RNA PCR testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection; f. A known history of HIV seropositivity; g. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection); h. Patients with an active, bleeding diathesis
11. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. Adequate contraception must be used throughout the trial and for 8 weeks after the last dose of study drug, by both sexes. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of everolimus)
12. Patients who have received prior treatment with an mTOR inhibitor (e.g., sirolimus, temsirolimus, everolimus).
13. Patients with a known hypersensitivity to everolimus or other rapamycins (e.g., sirolimus, temsirolimus) or to its excipients
14. History of noncompliance to medical regimens
15. Patients unwilling to or unable to comply with the protocol.
16. Patients with isolated recurrences (vaginal, pelvic, or paraaortic) that are amenable to potentially curative treatment with radiation therapy or surgery.
17. Patients with acute or chronic metabolic acidosis, lactic acidosis, or ketoacidosis. Note: during the study, metformin must be discontinued for 24 hours before and 48 hours after imaging involving IV contrast to minimize risk of lactic acidosis.
18. Patients who have hypoglycemia with a value of </= 50 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-10-07 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Rate (CBR) | 8 weeks
  Clinical benefit rate (CBR) determined by combining the complete response rate, partial response rate, and stable disease rate. Response evaluated by repeat imaging (CT or MRI) using RECIST 1.1 at the completion of the second cycle (8 weeks + 7 days of treatment).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 6 months
  Survival determined by measuring the time from study entry (1st treatment) to progression (PFS) or death (OS). Progression-free survival (PFS) and overall survival (OS) estimated with the Kaplan-Meier product-limit estimator.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Soliman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (6):
  - Sacred Heart Health Systems, Pensacola, Florida
  - MD Anderson Cooper Cancer Center, Voorhees Township, New Jersey
  - Memorial City Medical Center, Houston, Texas
  - Lyndon B Johnson General Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org